CLINICAL TRIAL: NCT04918342
Title: Comparison of Individualized Versus Group Telehealth Physical Therapy Programs for Individuals With Parkinson Disease
Brief Title: Group Versus Individuals Telehealth Exercise Programs for People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ithaca College (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 271
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either exercise individually with a physical therapist or in a group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Exercise Instruction (Active Comparator): The participant will receive individual exercise instruction.
  Interventions: Other: Multidimensional Exercise Program
- Group Exercise Instruction (Experimental): The participant will receive the instruction in a group of up to 9 other participants.
  Interventions: Other: Multidimensional Exercise Program

INTERVENTIONS:
Other: Multidimensional Exercise Program — The multidirectional exercise program will include cardiovascular training, strengthening, balance training, and flexibility training. This will be delivered 2 times per week for 8 weeks using telehealth and will be delivered by a physical therapist. The exercises will be modified to meet the participants needs. Intensity of exercise interventions will be monitored through patient self report and use of continuous heart rate monitoring.

SUMMARY:
This study will compare the impact of physical therapist led telehealth exercise programs on people with Parkinson disease. Eligible participants will complete this program individually or in a group of 9 other participants. The impact of participation in this program on motor function, postural control, gait, quality of life, and self-efficacy for exercise will be measured.

DETAILED DESCRIPTION:
This program will be delivered 2 times per week for 8 weeks with examination of outcome measures prior to and after completion. The investigators plan to enroll 20 participants with 10 completing a group program led by a physical therapist and 10 completing an individual exercise program led by a physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of idiopathic Parkinson disease
* been prescribed a stable dose of levadopa medication for at least 4 weeks prior to study participation
* be able to walk independently
* have a referral from a physician to participate in the program
* have access to a computer/tablet/or phone to use for telehealth sessions with reliable internet and access to the Zoom platform

Exclusion Criteria:

* have any other neurological condition other than Parkinson disease
* have a score less than 20/28 on the Mini-Balance Systems Evaluation Test (reflecting a higher risk of falls)
* demonstrate unstable/unsafe blood pressure or heart rate responses during the initial evaluation with response to submaximal exercise
* have any musculoskeletal condition that affected their ability to participate in the exercise group
* score less than 24/30 on the Mini Mental Status Examination during the initial evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in "Mini-Balance Evaluation Systems Test" Score | Prior to and after the 8 week intervention.
  This is a 14 item outcome measure that examines postural control in standing. The measure includes items that assess anticipatory postural control, reactive postural control, somatosensory integration, and dynamic gait. The scores range from 0-28 points with 28 reflecting the best possible balance performance.
Change in "Five Times Sit to Stand" test time | Prior to and after the 8 week intervention.
  For this outcome the participant is asked to perform sitting to standing transitions 5 times as quickly as possible. The time to complete the task is recorded. A lower time is associated with faster and more agile performance with sitting to standing transitions.

SECONDARY OUTCOMES:
Change in 10 meter walk test | Prior to and after 8 week intervention.
  This outcome measure examines gait speed at comfortable and fast speeds. This will be performed using the Gait Rite mat which will collect information about gait characteristics, including step length, step width, and gait symmetry as well. A faster time is associated with better balance and walking ability.
Change in Six Minute Walk Test Distance | Prior to and after 8 week intervention.
  This outcome examines gait endurance by measuring the distance walked over 6 minutes on a level surface. A greater number of meters on the test is associated with better walking endurance.
Change in Parkinson Disease Questionnaire-39 score | Prior to and after 8 week intervention.
  This is a self report quality of life measure designed for individuals with Parkinson disease. There are 8 subsections which can be reported individually and the score can be calculated as a summary score out of 100%. A lower percentage is associated with lower disability related to Parkinson disease.
Change in Self Efficacy for Exercise Scale score | Prior to and after 8 week intervention.
  This measures a person's confidence that they will exercise in a variety of situations.The score ranges from 0 to 90 with a higher score associated with a higher self efficacy for exercise behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fishel, Principal Investigator — Faculty
Locations (1):
- Sarah Fishel, Ithaca, New York, United States